CLINICAL TRIAL: NCT05944003
Title: Resuscitative Thoracotomy Practices
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 015.TRA.2022.D
Record Dates: First submitted 2023-07-06; First posted 2023-07-13 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Resuscitative Thoracotomy Practices

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Resuscitative thoracotomies — Resuscitative thoracotomies is an effective life saving measure in appropriate populations [1-8]. Unfortunately, when used outside of these populations the mortality rate is typically more than 90% [1-8]. Western Trauma Association and Eastern Association for the Surgery of Trauma have provided guidelines for which trauma patients are a candidate for RT [1-

SUMMARY:
Resuscitative thoracotomies (RT) are an effective life saving measure in appropriate populations [1-8]. Unfortunately, when used outside of these populations the mortality rate is typically more than 90% [1-8]. Western Trauma Association and Eastern Association for the Surgery of Trauma have provided guidelines for which trauma patients are a candidate for RT [1-3].

DETAILED DESCRIPTION:
EPIC and trauma registry will be queried for demographic information, admission dates, discharge diagnoses, inpatient cognitive function, routine testing (imaging and labs) reports, and surgical histories to determine number of patients who underwent RT, survived the RT, deficits from their cardiac arrest, and if they were COVID-19 positive. A full list of variables to be extracted from the chart review is in Appendix B. Chart review and data collection for these patients should be completed by December of 2024.

ELIGIBILITY:
Inclusion Criteria:

* Trauma patients who underwent RT in the emergency department (ED), operating room (OR), or intensive care unit (ICU) from January 1, 2017 to December 31, 2023.

Exclusion Criteria:

* Trauma patients who did not have a RT in the ED, OR, or ICU or were less than 16 years old from January 1, 2017 to December 31, 2023.

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Trauma patients who underwent RT in the emergency department (ED), operating room (OR), or intensive care unit (ICU) from January 1, 2017 to December 31, 2023.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-05-18 (Actual); Primary Completion 2024-05-18 (Estimated); Study Completion 2024-05-18 (Estimated)

PRIMARY OUTCOMES:
Total number of RT (before and during the COVID-19 pandemic) | 2 years
  Determine the rate of RT at MDMC. Particularly, if there was an increase during the COVID-19 pandemic, which would lead to greater exposure to transmissible disease

SECONDARY OUTCOMES:
• Cognitive deficits of any survivors of RT (GCS, assessments by neurology, mental status exams, and/or similar assessments documented in the EMR) | 2 yrs
  • Determine the rate of RT at MDMC. Particularly, if there was an increase during the COVID-19 pandemic, which would lead to greater exposure to transmissible disease

CONTACTS AND LOCATIONS:
Locations (1):
- Methodist Dallas Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Study data or any protected health information will not be shared with anyone that is not delegated to the study. The PI is committed to disseminate research results in a timely fashion. Sharing of results generated by the data analysis during the course of the project will be through presentation at national scientific meetings and/or publication in open access journals. All information obtained will be source de-identified and presented on a large scale and not traceable to any one particular individual.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: with in 1-2 years
Access Criteria: The data will be presented at local, regional, national, and international sites. The research gathered will be analyzed and submitted to relevant peer-reviewed medical journals for publication to add to the body of knowledge in the science community. Our potential list of conferences include: AAST (American Association for the Surgery of Trauma), SWSC (Southwest Surgical Congress), EAST (Eastern Association for the Surgery of Trauma), WTA (Western Trauma Association), or similar.

REFERENCES:
- [Background] Burlew CC, Moore EE, Moore FA, Coimbra R, McIntyre RC Jr, Davis JW, Sperry J, Biffl WL. Western Trauma Association critical decisions in trauma: resuscitative thoracotomy. J Trauma Acute Care Surg. 2012 Dec;73(6):1359-63. doi: 10.1097/TA.0b013e318270d2df. PMID 23188227
- [Background] Moore EE, Knudson MM, Burlew CC, Inaba K, Dicker RA, Biffl WL, Malhotra AK, Schreiber MA, Browder TD, Coimbra R, Gonzalez EA, Meredith JW, Livingston DH, Kaups KL; WTA Study Group. Defining the limits of resuscitative emergency department thoracotomy: a contemporary Western Trauma Association perspective. J Trauma. 2011 Feb;70(2):334-9. doi: 10.1097/TA.0b013e3182077c35. PMID 21307731
- [Background] Seamon MJ, Haut ER, Van Arendonk K, Barbosa RR, Chiu WC, Dente CJ, Fox N, Jawa RS, Khwaja K, Lee JK, Magnotti LJ, Mayglothling JA, McDonald AA, Rowell S, To KB, Falck-Ytter Y, Rhee P. An evidence-based approach to patient selection for emergency department thoracotomy: A practice management guideline from the Eastern Association for the Surgery of Trauma. J Trauma Acute Care Surg. 2015 Jul;79(1):159-73. doi: 10.1097/TA.0000000000000648. PMID 26091330
- [Background] Aseni P, Rizzetto F, Grande AM, Bini R, Sammartano F, Vezzulli F, Vertemati M. Emergency Department Resuscitative Thoracotomy: Indications, surgical procedure and outcome. A narrative review. Am J Surg. 2021 May;221(5):1082-1092. doi: 10.1016/j.amjsurg.2020.09.038. Epub 2020 Oct 2. PMID 33032791
- [Background] Hughes M, Perkins Z. Outcomes following resuscitative thoracotomy for abdominal exsanguination, a systematic review. Scand J Trauma Resusc Emerg Med. 2020 Feb 6;28(1):9. doi: 10.1186/s13049-020-0705-4. PMID 32028977
- [Background] Rhee PM, Acosta J, Bridgeman A, Wang D, Jordan M, Rich N. Survival after emergency department thoracotomy: review of published data from the past 25 years. J Am Coll Surg. 2000 Mar;190(3):288-98. doi: 10.1016/s1072-7515(99)00233-1. PMID 10703853
- [Background] Powell DW, Moore EE, Cothren CC, Ciesla DJ, Burch JM, Moore JB, Johnson JL. Is emergency department resuscitative thoracotomy futile care for the critically injured patient requiring prehospital cardiopulmonary resuscitation? J Am Coll Surg. 2004 Aug;199(2):211-5. doi: 10.1016/j.jamcollsurg.2004.04.004. PMID 15275875
- [Background] Panossian VS, Nederpelt CJ, El Hechi MW, Chang DC, Mendoza AE, Saillant NN, Velmahos GC, Kaafarani HMA. Emergency Resuscitative Thoracotomy: A Nationwide Analysis of Outcomes and Predictors of Futility. J Surg Res. 2020 Nov;255:486-494. doi: 10.1016/j.jss.2020.05.048. Epub 2020 Jul 1. PMID 32622163
- [Background] Inaba K, Chouliaras K, Zakaluzny S, Swadron S, Mailhot T, Seif D, Teixeira P, Sivrikoz E, Ives C, Barmparas G, Koronakis N, Demetriades D. FAST ultrasound examination as a predictor of outcomes after resuscitative thoracotomy: a prospective evaluation. Ann Surg. 2015 Sep;262(3):512-8; discussion 516-8. doi: 10.1097/SLA.0000000000001421. PMID 26258320
- [Background] Soreide K, Petrone P, Asensio JA. Emergency thoracotomy in trauma: rationale, risks, and realities. Scand J Surg. 2007;96(1):4-10. doi: 10.1177/145749690709600102. PMID 17461305